CLINICAL TRIAL: NCT04908722
Title: A Randomized, Double-blind, Phase 3 Study to Evaluate 6 Dose Levels of Ad26.COV2.S Administered As a Two-Dose Schedule in Healthy Adults
Brief Title: A Study to Evaluate Dose Levels of Ad26.COV2.S Administered as a Two-dose Schedule in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108960; 2020-005801-14 (EudraCT Number); VAC31518COV3003 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Prevention
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group 1: Ad26.COV2.S Dose Level 1 (Experimental): Participants in the main study and sub study will receive intramuscular (IM) injections of Ad26.COV2.S as a 2-dose vaccination regimen at dose level 1 on Days 1 and 57.
  Interventions: Biological: Ad26.COV2.S
- Group 2: Ad26.COV2.S Dose Level 2 (Experimental): Participants will receive IM injections of Ad26.COV2.S as a 2-dose vaccination regimen at dose level 2 on Days 1 and 57 in the main study.
  Interventions: Biological: Ad26.COV2.S
- Group 3: Ad26.COV2.S Dose Level 3 (Experimental): Participants in the main study and sub study will receive IM injections of Ad26.COV2.S as a 2-dose vaccination regimen at dose level 3 on Days 1 and 57.
  Interventions: Biological: Ad26.COV2.S
- Group 4: Ad26.COV2.S Dose Level 4 (Experimental): Participants will receive IM injections of Ad26.COV2.S as a 2-dose vaccination regimen at dose level 4 on Days 1 and 57 in the main study.
  Interventions: Biological: Ad26.COV2.S
- Group 5: Ad26.COV2.S Dose Level 5 (Experimental): Participants in the main study and sub study will receive IM injections of Ad26.COV2.S as a 2-dose vaccination regimen at dose level 5 on Days 1 and 57.
  Interventions: Biological: Ad26.COV2.S
- Group 6: Ad26.COV2.S Dose Level 6 (Experimental): Participants in the main study and sub study will receive IM injections of Ad26.COV2.S as a 2-dose vaccination regimen at dose level 6 on Days 1 and 57.
  Interventions: Biological: Ad26.COV2.S

INTERVENTIONS:
Biological: Ad26.COV2.S — Participants will receive intramuscular (IM) injections of Ad26.COV2.S.
  Other Names: JNJ-78436735; Ad26COVS1; VAC31518

SUMMARY:
The purpose of this study is to demonstrate non-inferiority (NI) in terms of humoral immune responses after 6 dose levels of Ad26.COV2.S.

ELIGIBILITY:
Inclusion Criteria:

* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study
* Participant must be healthy, in the investigator's clinical judgment, as confirmed by medical history, physical examination, and vital signs performed at screening. Participant may have underlying illnesses, as long as the symptoms and signs are medically controlled and not considered to be comorbidities related to an increased risk of severe Coronavirus disease 2019 (COVID-19), except for smoking, which is allowed. If on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participant will be included on the basis of physical examination, medical history, and vital signs
* All female participants of childbearing potential must: a) have a negative highly sensitive urine pregnancy test at screening; b) have a negative highly sensitive urine pregnancy test immediately prior to each study vaccine administration
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine
* Participant must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius (C) (100.4 degree Fahrenheit [F]) within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Participant received or plans to receive: (a) licensed live attenuated vaccines - within 28 days before or after planned administration of the first or subsequent study vaccinations; and (b) other licensed (not live) vaccines - within 14 days before or after planned administration of the first or subsequent study vaccinations
* Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) or used an invasive investigational medical device within 30 days or received investigational immunoglobulin (Ig) or monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine within 6 months before the planned administration of the first dose of study vaccine or is currently enrolled or plans to participate in another investigational study during the course of this study
* Participant previously received a coronavirus vaccine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1609 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (43):
- United States (18):
  - Baptist Health Center For Clinical Research, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Ark Clinical Research, Long Beach, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - Wr McCr Llc, San Diego, California
  - Ark Clinical Research, Tustin, California
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Floridian Research Institute, Miami, Florida
  - Medpharmics, LLC, Metairie, Louisiana
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Rochester Clinical Research, Inc, Rochester, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Tekton Research Inc., Yukon, Oklahoma
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Ventavia Research Group, LLC, Keller, Texas
  - Research Your Health, Plano, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia
- Brazil (11):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - CECOR Centro OncolOgico de Roraima, Boa Vista
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - Núcleo de Medicina Tropical - Universidade Federal do Ceará, Ceará
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas - CEPCLIN, Natal
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Municipio de Nova Iguacu - Hospital Geral de Nova Iguacu, Rio de Janeiro
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - Centro de Referencia E Treinamento Dst/Aids, São Paulo
- Germany (5):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Clinical Research HamburggmbH, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Synexus Clinical Research GmbH, Leipzig
  - Universitaetsmedizin Rostock, Rostock
- Poland (3):
  - Gdanskie Centrum Zdrowia, Gdansk
  - Centrum Medyczne Medyk, Rzeszów
  - Centrum Medyczne Pratia Poznan, Skorzewo
- South Africa (6):
  - Synexus Helderberg Clinical Research Centre, Cape Town
  - Ndlovu Elandsdoorn Site, Dennilton
  - Stanza Clinical Research Centre : Mamelodi, Mamelodi East
  - PHOENIX PHARMA (Pty) Ltd, Port Elizabeth
  - Gct Sunnyside, Pretoria
  - Setshaba Research Centre, Soshanguve

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1609 participants were enrolled, but 1 participant was randomized by error. This participant was never treated and was removed from the randomized list.
Pre-assignment Details: As planned, the Participant flow, baseline characteristics, Outcome measures data and adverse events data were analyzed and reported combined for the main study and sub-study.
Groups:
- Group 1: Ad26.COV2.S 9x10^10 vp: Participants in the main study and sub study received Intramuscular (IM) injection of Ad26.COV2.S 9x10^10 viral particles (vp) on Days 1 and 57.
- Group 2: Ad26.COV2.S 7x10^10 vp: Participants in the main study received IM injection of Ad26.COV2.S 7x10^10 vp on Days 1 and 57.
- Group 3: Ad26.COV2.S 5x10^10 vp: Participants in the main study and sub study received IM injection of Ad26.COV2.S 5x10^10 vp on Days 1 and 57.
- Group 4: Ad26.COV2.S 3.5x10^10 vp: Participants in the main study received IM injection of Ad26.COV2.S 3.5x10^10 vp on Days 1 and 57.
- Group 5: Ad26.COV2.S 2.5x10^10 vp: Participants in the main study and sub study received IM injection of Ad26.COV2.S 2.5x10^10 vp on Days 1 and 57.
- Group 6: Ad26.COV2.S 1.25x10^10 vp: Participants in the main study and sub study received IM injection of Ad26.COV2.S 1.25x10^10 vp on Days 1 and 57.
Period: Overall Study
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Started (Randomized Participants) | 291 | 222 | 293 | 222 | 291 | 289
Main Study | 222 | 222 (Participants in Group 2 were not enrolled in the sub-study.) | 223 | 222 (Participants in Group 4 were not enrolled in the sub-study.) | 222 | 221
Sub Study | 69 | 0 (Participants in Group 2 were not enrolled in the sub-study.) | 70 | 0 (Participants in Group 4 were not enrolled in the sub-study.) | 69 | 68
Treated (Vaccinated Participants) | 288 | 221 | 291 | 220 | 288 | 285
Per Protocol Immunogenicity Set | 276 | 212 | 282 | 212 | 277 | 271
Completed | 237 | 178 | 244 | 179 | 240 | 233
Not Completed | 54 | 44 | 49 | 43 | 51 | 56
Not completed — Protocol deviation | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 33 | 33 | 36 | 30 | 32 | 34
Not completed — Physician Decision | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 8 | 7 | 6 | 12 | 14
Not completed — Other | 3 | 1 | 3 | 2 | 4 | 1
Not completed — Initiated prohibited medication | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Randomized but not vaccinated | 3 | 1 | 2 | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants with at least one vaccine administration documented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp | Total
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285 | 1593
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.21) | 35.2 (9.87) | 34.8 (9.82) | 34.7 (9.36) | 34.5 (9.81) | 33.4 (9.63) | 34.7 (9.81)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 288 | 221 | 291 | 220 | 288 | 285 | 1593
  From 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 117 | 73 | 119 | 72 | 106 | 103 | 590
  Male | 170 | 148 | 172 | 148 | 182 | 182 | 1002
  Undifferentiated | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 132 | 83 | 129 | 87 | 121 | 130 | 682
  Not Hispanic or Latino | 130 | 123 | 138 | 116 | 137 | 135 | 779
  Unknown or Not Reported | 26 | 15 | 24 | 17 | 30 | 20 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 1 | 0 | 0 | 6
  Asian | 3 | 3 | 4 | 3 | 2 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Black or African American | 104 | 57 | 90 | 63 | 87 | 101 | 502
  White | 161 | 142 | 174 | 138 | 183 | 163 | 961
  More than one race | 2 | 1 | 4 | 4 | 3 | 2 | 16
  Unknown or Not Reported | 16 | 17 | 15 | 11 | 12 | 15 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 155 | 112 | 152 | 104 | 146 | 142 | 811
  Germany | 56 | 59 | 64 | 65 | 59 | 65 | 368
  South Africa | 22 | 14 | 25 | 13 | 24 | 24 | 122
  United States | 55 | 36 | 50 | 38 | 59 | 54 | 292

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) S Protein Binding Antibodies Measured by Enzyme-Linked Immunosorbent Assay (ELISA) 28 Days After First Vaccination
Description: Geometric mean concentration of SARS-CoV-2 S protein binding antibodies measured by ELISA were reported. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: 28 days after first vaccination (at Day 29)
Population: The per protocol immunogenicity set included all randomized and vaccinated participants for whom immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, 'N' (number of participants analysed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per millilitre (EU/mL)
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 249 | 191 | 250 | 189 | 243 | 251
ELISA Units per millilitre (EU/mL) | 2351 [1849 to 2989] | 1714 [1305 to 2250] | 2189 [1726 to 2775] | 1377 [1062 to 1786] | 1626 [1255 to 2106] | 1976 [1521 to 2566]
Statistical Analysis 1: Comparison: Group 1: Ad26.COV2.S 9x10^10 vp vs Group 3: Ad26.COV2.S 5x10^10 vp; Group 1 (1 dose) vs Group 3 (1 dose); Test type: Non-Inferiority — Tested using 97.5% confidence interval approach. The non-inferiority margin was 0.67; Geometric mean ratio = 1.15, 97.5% CI 2-sided [0.926 to 1.440]
Statistical Analysis 2: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 5: Ad26.COV2.S 2.5x10^10 vp; Group 5 (1 dose) vs Group 3 (1 dose); Test type: Non-Inferiority — Tested using 97.5% confidence interval approach. The non-inferiority margin was 0.67; Geometric mean ratio = 0.80, 97.5% CI [0.641 to 1.00]
Statistical Analysis 3: Comparison: Group 2: Ad26.COV2.S 7x10^10 vp vs Group 3: Ad26.COV2.S 5x10^10 vp; Group 2 (1 dose) vs Group 3 (1 dose); Test type: Non-Inferiority — Tested using 97.5% confidence interval approach. The non-inferiority margin was 0.67; Geometric mean ratio = 1.07, 97.5% CI 2-sided [0.844 to 1.356]
Statistical Analysis 4: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 4: Ad26.COV2.S 3.5x10^10 vp; Group 4 (1 dose) vs Group 3 (1 dose); Test type: Non-Inferiority — Tested using 97.5% confidence interval approach. The non-inferiority margin was 0.67; Geometric mean ratio = 0.94, 97.5% CI 2-sided [0.742 to 1.193]
Statistical Analysis 5: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 6: Ad26.COV2.S 1.25x10^10 vp; Group 6 (1 dose) vs Group 3 (1 dose); Test type: Non-Inferiority — Tested using 97.5% confidence interval approach. The non-inferiority margin was 0.67; Geometric mean ratio = 0.81, 97.5% CI 2-sided [0.648 to 1.007]

2. Primary Outcome: Geometric Mean Concentration of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) S Protein Binding Antibodies Measured by Enzyme-Linked Immunosorbent Assay (ELISA) 14 Days After Second Vaccination
Description: as for outcome 1
Time Frame: 14 days after second vaccination (at Day 71)
Population: The per protocol immunogenicity set included all randomized and vaccinated participants for whom immunogenicity data were available excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per millilitre (EU/mL)
Groups:
- Group 4: Ad26.COV2.S 3.5x10^10 vp: Participants in the main study received IM injection of Ad26.COV2.S 3.5x10^10 vp on Days 1 and Day 57.
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 171 | 130 | 180 | 134 | 172 | 184
ELISA Units per millilitre (EU/mL) | 4997 [4145 to 6023] | 3757 [3030 to 4659] | 3855 [3185 to 4666] | 3460 [2781 to 4304] | 3641 [2969 to 4465] | 3905 [3113 to 4897]
Statistical Analysis 1: Comparison: Group 1: Ad26.COV2.S 9x10^10 vp vs Group 3: Ad26.COV2.S 5x10^10 vp; Group 1 (2 doses) vs Group 3 (1 dose); Test type: Non-Inferiority — Testing according to sequential non-inferiority assessment hypothesis. Tested using 97.5% confidence interval approach. The non-inferiority margin was 0.67; Geometric mean ratio = 2.53, 97.5% CI 2-sided [1.992 to 3.207]
Statistical Analysis 2: Comparison: Group 1: Ad26.COV2.S 9x10^10 vp vs Group 3: Ad26.COV2.S 5x10^10 vp; Group 1 (2 doses) vs Group 3 (2 doses); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 1.41, 97.5% CI 2-sided [1.088 to 1.815]
Statistical Analysis 3: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 5: Ad26.COV2.S 2.5x10^10 vp; Group 5 (2 doses) vs Group 3 (1 dose); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 1.79, 97.5% CI 2-sided [1.408 to 2.265]
Statistical Analysis 4: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 5: Ad26.COV2.S 2.5x10^10 vp; Group 5 (2 doses) vs Group 3 (2 doses); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.99, 97.5% CI 2-sided [0.769 to 1.282]
Statistical Analysis 5: Comparison: Group 2: Ad26.COV2.S 7x10^10 vp vs Group 3: Ad26.COV2.S 5x10^10 vp; Group 2 (2 doses) vs Group 3 (1 dose); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 2.37, 97.5% CI 2-sided [1.829 to 3.007]
Statistical Analysis 6: Comparison: Group 2: Ad26.COV2.S 7x10^10 vp vs Group 3: Ad26.COV2.S 5x10^10 vp; Group 2 (2 doses) vs Group 3 (2 doses); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 1.32, 97.5% CI 2-sided [1.000 to 1.739]
Statistical Analysis 7: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 4: Ad26.COV2.S 3.5x10^10 vp; Group 4 (2 doses) vs Group 3 (1 dose); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 2.20, 97.5% CI 2-sided [1.697 to 2.841]
Statistical Analysis 8: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 4: Ad26.COV2.S 3.5x10^10 vp; Group 4 (2 doses) vs Group 3 (2 doses); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 1.22, 97.5% CI 2-sided [0.928 to 1.606]
Statistical Analysis 9: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 6: Ad26.COV2.S 1.25x10^10 vp; Group 6 (2 doses) vs Group 3 (1 dose); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 1.70, 97.5% CI 2-sided [1.348 to 2.148]
Statistical Analysis 10: Comparison: Group 3: Ad26.COV2.S 5x10^10 vp vs Group 6: Ad26.COV2.S 1.25x10^10 vp; Group 6 (2 doses) vs Group 3 (2 doses); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Geometric mean ratio = 0.95, 97.5% CI 2-sided [0.736 to 1.217]

3. Secondary Outcome: Percentage of Participants With Serological Response to Vaccination to SARS-COV-2 S Protein as Measured by ELISA
Description: Percentage of participants with serological response to vaccination to SARS-COV-2 S protein as measured by ELISA were reported. A participant was considered a responder if one or both of the following conditions were satisfied: (1) the baseline (pre-dose 1) sample value was less than or equal to (<=) lower limit of quantification (LLOQ) and the post-baseline sample was greater than (>) LLOQ; (2) the baseline sample (pre-dose 1) value was >LLOQ and the post-baseline sample value represented an at least 4-fold (>=4-fold) increase from the baseline sample value. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: Day 29, Day 57, Day 71, Week 32, and Week 60
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 249 | 191 | 250 | 189 | 243 | 251
Percentage of participants
  Day 29 | 82.7 | 90.1 | 78.8 | 87.8 | 80.2 | 76.1
  Day 57: number analyzed (Participants) | 216 | 167 | 217 | 162 | 219 | 220
  Day 57 | 81.9 | 88.6 | 80.2 | 92.0 | 81.3 | 77.7
  Day 71: number analyzed (Participants) | 171 | 130 | 180 | 134 | 172 | 184
  Day 71 | 81.9 | 92.3 | 79.4 | 91.8 | 80.8 | 76.1
  Week 32: number analyzed (Participants) | 112 | 86 | 128 | 90 | 121 | 136
  Week 32 | 72.3 | 83.7 | 68.0 | 86.7 | 68.6 | 63.2
  Week 60: number analyzed (Participants) | 45 | 33 | 42 | 37 | 45 | 52
  Week 60 | 68.9 | 81.8 | 61.9 | 83.8 | 60.0 | 53.8

4. Secondary Outcome: Geometric Mean Concentration of SARS-CoV-2 S Protein Binding Antibody Measured by ELISA
Description: Geometric mean concentration of SARS-CoV-2 S protein binding antibody measured by ELISA were reported. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: Day 29, Day 57, Day 71, Week 32, and Week 60
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Unit (EU)/mL
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 249 | 191 | 250 | 189 | 243 | 251
ELISA Unit (EU)/mL
  Day 29 | 2351 [1849 to 2989] | 1714 [1305 to 2250] | 2189 [1726 to 2775] | 1377 [1062 to 1786] | 1626 [1255 to 2106] | 1976 [1521 to 2566]
  Day 57: number analyzed (Participants) | 216 | 167 | 217 | 162 | 219 | 220
  Day 57 | 2722 [2156 to 3438] | 1842 [1404 to 2417] | 2089 [1651 to 2643] | 1622 [1233 to 2134] | 1919 [1481 to 2486] | 2293 [1766 to 2978]
  Day 71: number analyzed (Participants) | 171 | 130 | 180 | 134 | 172 | 184
  Day 71 | 4997 [4145 to 6023] | 3757 [3030 to 4659] | 3855 [3185 to 4666] | 3460 [2781 to 4304] | 3641 [2969 to 4465] | 3905 [3113 to 4897]
  Week 32: number analyzed (Participants) | 112 | 86 | 128 | 90 | 121 | 136
  Week 32 | 3331 [2499 to 4438] | 2903 [2076 to 4058] | 2616 [2001 to 3420] | 2059 [1470 to 2885] | 3067 [2268 to 4148] | 2707 [2000 to 3662]
  Week 60: number analyzed (Participants) | 45 | 33 | 42 | 37 | 45 | 52
  Week 60 | 4968 [3119 to 7915] | 5010 [3146 to 7981] | 2363 [1448 to 3857] | 2191 [1224 to 3921] | 2769 [1776 to 4317] | 3664 [2169 to 6190]

5. Secondary Outcome: Number of Subjects With Solicited Local Adverse Events (AEs) for 7 Days After Each Vaccination
Description: An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participant in their e-diary for 7 days after each vaccination. Solicited local AEs included injection site pain/tenderness, erythema and swelling at the study vaccine injection site. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: 7 days after each vaccination (first vaccination [at Day 8], second vaccination [at Day 64])
Population: Full analysis set included all participants with at least one vaccine administration documented. Here, 'n' (number of participants analyzed) signifies number of participants evaluable for this timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants
  After first vaccination | 179 | 143 | 162 | 137 | 155 | 133
  After second vaccination: number analyzed (Participants) | 264 | 200 | 269 | 199 | 270 | 258
  After second vaccination | 130 | 100 | 124 | 95 | 111 | 104

6. Secondary Outcome: Number of Subjects With Solicited Systemic AEs for 7 Days After Each Vaccination
Description: An AE was any untoward medical occurrence in a subject participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited systemic AEs (include body temperature, fatigue, headache, nausea, myalgia) were noted in the subject diary after 7 days of each vaccination. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: 7 days after each vaccination (first vaccination [at Day 8], second vaccination [at Day 64])
Population: Full analysis set included all participants with at least one vaccine administration documented. Here, 'n' (number of subjects analysed) signifies number of subjects evaluable for this timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants
  After first vaccination | 204 | 156 | 173 | 135 | 156 | 152
  After second vaccination: number analyzed (Participants) | 264 | 200 | 269 | 199 | 270 | 258
  After second vaccination | 144 | 98 | 111 | 91 | 105 | 109

7. Secondary Outcome: Number of Participants With Unsolicited AEs for 28 Days After Each Vaccination
Description: Unsolicited AEs were all AEs for which the subject was not specifically questioned in the subject diary. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: 28 days after each vaccination (first vaccination [at Day 29], second vaccination [at Day 85])
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants
  After first vaccination | 78 | 60 | 55 | 58 | 69 | 59
  After second vaccination: number analyzed (Participants) | 264 | 200 | 269 | 199 | 270 | 258
  After second vaccination | 55 | 28 | 49 | 39 | 53 | 50

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE was any untoward medical occurrence that at any dose may results in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: From Day 1 (post-vaccination) up to end of the study (up to 60 weeks)
Population: Full analysis set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants | 13 | 3 | 4 | 4 | 3 | 5

9. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with thrombocytopenia syndrome were considered to be an AESI. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: From Day 1 (post-vaccination) up to end of the study (up to 60 weeks)
Population: Full analysis set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With AEs Leading to Study Discontinuation
Description: Number of participants with AEs leading to study discontinuation were reported. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: Up to 60 weeks
Population: Full analysis set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Ad26.COV2.S 9x10^10 vp: Participants in the main study received Intramuscular (IM) injection of Ad26.COV2.S 9x10^10 viral particles (vp) on Days 1 and 57.
- Group 3: Ad26.COV2.S 5x10^10 vp: Participants in the main study received IM injection of Ad26.COV2.S 5x10^10 vp on Days 1 and 57.
- Group 5: Ad26.COV2.S 2.5x10^10 vp: Participants in the main study received IM injection of Ad26.COV2.S 2.5x10^10 vp on Days 1 and 57.
- Group 6: Ad26.COV2.S 1.25x10^10 vp: Participants in the main study received IM injection of Ad26.COV2.S 1.25x10^10 vp on Days 1 and 57.
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Medically-Attended Adverse Events (MAAEs)
Description: MAAEs were defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits were not considered medically-attended visits. New onset of chronic diseases were collected as part of the MAAEs. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Time Frame: 6 months after second vaccination (up to 32 weeks)
Population: Full analysis set included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
Number analyzed (Participants) | 288 | 221 | 291 | 220 | 288 | 285
Participants | 54 | 34 | 50 | 35 | 48 | 35

ADVERSE EVENTS:
Time Frame: From Day 1 (post-vaccination) up to end of the study (up to 60 weeks)
Description: Full analysis set included all participants with at least one vaccine administration documented. As per planned analysis, the data were analyzed and reported combined for the main study and sub-study.
Arm/Group | Group 1: Ad26.COV2.S 9x10^10 vp | Group 2: Ad26.COV2.S 7x10^10 vp | Group 3: Ad26.COV2.S 5x10^10 vp | Group 4: Ad26.COV2.S 3.5x10^10 vp | Group 5: Ad26.COV2.S 2.5x10^10 vp | Group 6: Ad26.COV2.S 1.25x10^10 vp
All-Cause Mortality (participants affected / at risk) | 1/288 | 0/221 | 0/291 | 0/220 | 0/288 | 1/285
Serious Adverse Events (participants affected / at risk) | 13/288 | 3/221 | 4/291 | 4/220 | 3/288 | 5/285
Other Adverse Events (participants affected / at risk) | 245/288 | 187/221 | 236/291 | 188/220 | 228/288 | 217/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.COV2.S 9x10^10 vp (N=288) | Group 2: Ad26.COV2.S 7x10^10 vp (N=221) | Group 3: Ad26.COV2.S 5x10^10 vp (N=291) | Group 4: Ad26.COV2.S 3.5x10^10 vp (N=220) | Group 5: Ad26.COV2.S 2.5x10^10 vp (N=288) | Group 6: Ad26.COV2.S 1.25x10^10 vp (N=285)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid Artery Dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myasthenia Gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian Disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.COV2.S 9x10^10 vp (N=288) | Group 2: Ad26.COV2.S 7x10^10 vp (N=221) | Group 3: Ad26.COV2.S 5x10^10 vp (N=291) | Group 4: Ad26.COV2.S 3.5x10^10 vp (N=220) | Group 5: Ad26.COV2.S 2.5x10^10 vp (N=288) | Group 6: Ad26.COV2.S 1.25x10^10 vp (N=285)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 8 (9) | 0 (0) | 6 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 5 (6) | 1 (1) | 7 (8) | 4 (5) | 9 (15)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (3) | 3 (4) | 3 (5) | 2 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (6) | 2 (2) | 5 (5) | 5 (5) | 5 (6)
Nausea(Solicited) (Gastrointestinal disorders) | 95 (123) | 78 (99) | 67 (79) | 58 (71) | 64 (78) | 65 (80)
Odynophagia (Gastrointestinal disorders) | 3 (3) | 5 (7) | 3 (3) | 1 (1) | 2 (3) | 5 (7)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 2 (3)
Chills (General disorders) | 11 (13) | 5 (5) | 2 (2) | 5 (6) | 4 (4) | 0 (0)
Fatigue (General disorders) | 15 (19) | 11 (14) | 7 (9) | 9 (9) | 5 (5) | 15 (22)
Fatigue(Solicited) (General disorders) | 171 (248) | 140 (202) | 144 (207) | 113 (164) | 124 (173) | 132 (178)
Pyrexia (General disorders) | 9 (14) | 10 (14) | 5 (7) | 4 (4) | 4 (4) | 7 (7)
Pyrexia(Solicited) (General disorders) | 68 (77) | 41 (42) | 33 (37) | 27 (27) | 22 (25) | 16 (17)
Vaccination Site Erythema(Solicited) (General disorders) | 3 (3) | 5 (5) | 9 (9) | 4 (4) | 2 (2) | 5 (5)
Vaccination Site Pain (General disorders) | 7 (8) | 8 (12) | 4 (6) | 3 (4) | 6 (6) | 8 (10)
Vaccination Site Pain(Solicited) (General disorders) | 198 (306) | 156 (242) | 190 (284) | 153 (231) | 175 (265) | 160 (234)
Vaccination Site Swelling(Solicited) (General disorders) | 8 (8) | 9 (9) | 9 (12) | 3 (3) | 3 (3) | 8 (9)
Covid-19 (Infections and infestations) | 9 (14) | 21 (30) | 20 (28) | 20 (29) | 22 (35) | 13 (19)
Influenza (Infections and infestations) | 35 (57) | 26 (31) | 38 (50) | 26 (41) | 37 (52) | 25 (35)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7) | 7 (8) | 6 (8) | 8 (13) | 12 (13)
Rhinitis (Infections and infestations) | 8 (9) | 6 (8) | 1 (2) | 4 (4) | 10 (11) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 12 (17) | 6 (8) | 12 (15) | 7 (7) | 18 (20)
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 183 (260) | 126 (175) | 144 (188) | 115 (159) | 118 (159) | 111 (151)
Headache (Nervous system disorders) | 26 (28) | 14 (20) | 11 (12) | 21 (25) | 23 (26) | 22 (28)
Headache(Solicited) (Nervous system disorders) | 184 (260) | 139 (202) | 146 (195) | 109 (150) | 133 (175) | 123 (165)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (7) | 3 (4) | 7 (7) | 7 (8) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 2 (3) | 1 (2) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 6 (9) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT04908722/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT04908722/SAP_001.pdf